CLINICAL TRIAL: NCT05401591
Title: Microalgae as an Alternative Protein Source in Human Nutrition.
Acronym: MAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 21-07-14-A-01
Record Dates: First submitted 2022-05-26; First posted 2022-06-02 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Milk protein (Active Comparator)
  Interventions: Dietary Supplement: Protein shake
- Whole cell chlorella (Experimental)
  Interventions: Dietary Supplement: Protein shake
- Cracked cell chlorella (Experimental)
  Interventions: Dietary Supplement: Protein shake
- Spirulina (Experimental)
  Interventions: Dietary Supplement: Protein shake

INTERVENTIONS:
Dietary Supplement: Protein shake — Participant will drink a protein shake made using each of the four protein types.

SUMMARY:
Protein is an essential part of the human diet. But with a growing global population and climate emergency, current sources of dietary protein are unable to continue to sustainably meet the global demand. To ensure future food security, new sustainable protein sources are required. Microalgae - a group of plant-like single cells - are thought to be a good option due to their sustainable farming methods and naturally high protein content. Long term health benefits of eating microalgae have been seen in humans. However, the time directly following microalgae ingestion has not been well studied but is an important period when considering a protein source. This research will compare the period after ingestion of three preparations and/or types of microalgae to a traditional source of protein.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 -30 kg/m2
* age 18 - 40 years
* healthy
* non-smoker

Exclusion Criteria:

* BMI <18.5 or >30 kg/m2
* smoker
* metabolic disease
* relevant food intolerance
* using medications known to affect metabolism

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Plasma amino acids | 5 hours postprandial
  Amino acid concentrations measured in participant plasma following the ingestion of protein drinks.

CONTACTS AND LOCATIONS:
Locations (1):
- Exeter University, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No